CLINICAL TRIAL: NCT00568633
Title: A California Cooperative Clinical Study Comparing Allogeneic Hematopoietic Cell Transplantation Using Nonmyeloablative Host Conditioning With Total Lymphoid Irradiation and Anti-thymocyte Globulin Versus Best Standard of Care in Acute Myeloid Leukemia (AML) in First Complete Remission
Brief Title: Allogeneic HCT Using Nonmyeloablative Host Conditioning With TLI & ATG vs SOC in AML
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Stanford University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Robert Lowsky, Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-05567; 97843 (Other: Stanford University Alternate IRB Approval Number); BMT190 (Other: OnCore)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Leukemia, Myeloid; Leukemia; Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia; Leukemia, Myeloid, Acute | interventions — Hematopoietic Stem Cell Transplantation; Transplantation; Antilymphocyte Serum; thymoglobulin; Cyclosporine; Mycophenolic Acid; Methylprednisolone Hemisuccinate; Methylprednisolone; Methylprednisolone Acetate; Standard of Care

STUDY DESIGN:
Intervention Model Description: Treatment assignment was based on availability of an HLA-matched donor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allo-HSCT + TLI + ATG (Experimental): Participants achieving complete remission after consolidation therapy & who have 5 of 6 HLA-match sibling donor to provide PBSC harvest for transplant. Pre-transplant subjects receive:
  * Total lymphoid radiation (TLI) Days -11 to -7, and Days -4 to -1 (2 fractions on day -1)
  * Anti-thymocyte globulin (ATG) Days -11 to -7
  * Methylprednisolone Days -11 to -7
  * Cyclosporine (CSP) Days -4 to +2
  * 5+ of 6 HLA-matched CD34+ cells on Day 0
  * Mycophenolate mofetil (MMF), Day 0 to Day +28
  Interventions: Procedure: Allogeneic HSCT; Drug: Anti-thymocyte globulin (ATG); Drug: Cyclosporine (CSP); Drug: Mycophenolate mofetil (MMF); Radiation: Total lymphoid irradiation (TLI); Drug: Methylprednisolone sodium succinate
- Best Standard Care (Active Comparator): Regular medical care for participants who achieve complete remission after standard consolidation therapy, but do not have a 5 of 6 HLA-match sibling donor. Treatment may consist of:
  * Additional consolidation chemotherapy (3-4 cycles of cytarabine +/- an anthracycline agent, or other consolidation)
  * Autologous transplantation
  * Non-Myeloablative unrelated-donor transplant, +/- TLI and ATG conditioning
  * Umbilical cord blood transplantation
  * Haploidentical transplantation
  Interventions: Drug: Best standard care

INTERVENTIONS:
Procedure: Allogeneic HSCT — Allogeneic, 5+ of 6 HLA-matched PBSC transplant from sibling, mobilized to target of 5 x 10e6 CD34+ cells/kg and < 7 x 10e8 CD3+ cells/kg.
  Other Names: Hematopoietic stem cell transplantation (HSCT); Peripheral blood stem cell (PBSC) transplantation
  Arms: Allo-HSCT + TLI + ATG
Drug: Anti-thymocyte globulin (ATG) — 1.5 mg/kg for 5 days by IV
  Other Names: Thymoglobulin; Anti-thymocyte globulin (rabbit) (ATG)
  Arms: Allo-HSCT + TLI + ATG
Drug: Cyclosporine (CSP) — 6.25 mg/kg twice daily oral
  Other Names: Ciclosporin; cyclosporin A; cyclosporin
  Arms: Allo-HSCT + TLI + ATG
Drug: Mycophenolate mofetil (MMF) — 15 mg/kg twice daily oral
  Other Names: Cellcept
  Arms: Allo-HSCT + TLI + ATG
Radiation: Total lymphoid irradiation (TLI) — 80 cGy/fraction radiotherapy in 10 fractions.
  Arms: Allo-HSCT + TLI + ATG
Drug: Methylprednisolone sodium succinate — 1.0 mg/kg for 5 days by IV
  Other Names: Solumedrol; Medrol; Depo-Medrol; P-Care D40; P-Care D80
  Arms: Allo-HSCT + TLI + ATG
Drug: Best standard care — Intervention consist of:
  * Consolidation chemotherapy (3-4 cycles of cytarabine +/- an anthracycline agent, or other consolidation)
  * Autologous transplantation
  * Non-Myeloablative unrelated-donor transplant, +/- TLI and ATG conditioning
  * Umbilical cord blood transplantation
  * Haploidentical transplantation
  Other Names: Standard of Care (physician discretion); Regular medical care
  Arms: Best Standard Care

SUMMARY:
Acute myeloid leukemia (AML) is a cancer of the bone marrow that mostly affects older adults. Even with the best chemotherapy, two-year disease-free survival is achieved in a minority of patients. Bone marrow transplantation from a sibling donor may improve cure rates; however, patients over 50 years of age have a high risk of complications and therefore generally are excluded from this treatment option. Recently our group developed a transplantation strategy for older cancer patients that protects against transplant-associated complications, yet does not interfere with the ability of the transplanted donor cells to destroy cancer cells. With this new method, we can now safely evaluate transplantation as a curative therapy for AML patients over the age of 50. We have assembled clinical and scientific researchers throughout the state of California to study and compare bone marrow transplantation using our new approach with the best standard of care chemotherapy in AML patients over the age of 50. The results of this study have the potential to establish a new treatment standard that will improve survival of older AML patients.

ELIGIBILITY:
INCLUSION CRITERIA

* ≥ 50 years of age and ≤ 75 years of age.
* De novo acute myelogenous leukemia (AML), based on FAB and WHO criteria.
* Intermediate or unfavorable cytogenetic abnormalities based on Southwest Oncology Group (SWOG) Cytogenetic Criteria.
* First morphologic complete remission (CR), or CRp (a complete remission but with low platelets) following 1 or 2 courses of induction therapy, documented no more than 8 weeks prior to the date of enrollment and confirmed at time of enrollment.
* Karnofsky Performance Score ≥ 60.
* Suitable for non-myeloablative transplantation or best treatment.
* Able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA

* AML with favorable cytogenetic features based on SWOG Cytogenetic Criteria
* AML, either treatment-related or MDS-related
* Active CNS disease as identified by positive CSF cytospin at time of enrollment.
* Prior or concurrent malignancies except localized non-melanoma skin malignancies or treated cervical carcinoma in situ. (EXCEPTION: Cancer treated with curative intent > 5 years previously is allowed. EXCEPTION: Low grade lymphoma is allowed as long as active treatment is not required for control of disease)
* Planned for allogeneic transplant using a full-dose conditioning
* Life expectancy < 1 year due to diseases other than malignancy
* Pregnant or breastfeeding.
* HIV-seropositive.
* Uncontrolled infection (presumed or documented) with progression after appropriate therapy for greater than one month.
* Symptomatic coronary artery disease or uncontrolled congestive heart failure. Left ventricular ejection fraction (LVEF) is not required to be measured, however if measured, exclusion if ejection fraction is < 30%.
* Requiring supplementary continuous oxygen. Diffusing capacity of the lungs for carbon monoxide (DLCO) is not required to be measured, however if it is measured, exclusion if DLCO < 35%.
* Fulminant liver failure
* Cirrhosis with evidence of portal hypertension or bridging fibrosis
* Alcoholic hepatitis
* Esophageal varices
* A history of bleeding esophageal varices
* Hepatic encephalopathy
* Uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time
* Ascites related to portal hypertension
* Chronic viral hepatitis with total serum bilirubin > 3 mg/dL
* Symptomatic biliary disease

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - Kaiser Permanente Northern California, Hayward, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Univeristy of California Davis Medical Center, Sacramento, California
  - Stanford University School of Medicine, Stanford, California
  - West Virginia University Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Allo-HSCT + TLI + ATG: Participants achieving complete remission after consolidation therapy & who have 5 of 6 HLA-match sibling donor to provide PBSC harvest for transplant. Pre-transplant subjects receive:
  * Total lymphoid radiation (TLI) Days -11 to -7, and Days -4 to -1 (2 fractions on day -1)
  * Anti-thymocyte globulin (ATG) Days -11 to -7
  * Methylprednisolone Days -11 to -7
  * Cyclosporine (CSP) Days -4 to +2
  * 5+ of 6 HLA-matched CD34+ cells on Day 0
  * Mycophenolate mofetil (MMF), Day 0 to Day +28
  Allogeneic HSCT: Allogeneic, 5+ of 6 HLA-matched PBSC transplant from sibling, mobilized to target of 5 x 10e6 CD34+ cells/kg and < 7 x 10e8 CD3+ cells/kg.
  Anti-thymocyte globulin (ATG): 1.5 mg/kg for 5 days by IV
  Cyclosporine (CSP): 6.25 mg/kg twice daily oral
  Mycophenolate mofetil (MMF): 15 mg/kg twice daily oral
  Total lymphoid irradiation (TLI): 80 cGy/fraction radiotherapy in 10 fractions.
  Methylprednisolone sodium succinate: 1.0 mg/kg for 5 days by IV
- Best Standard Care: Regular medical care for participants who achieve complete remission after standard consolidation therapy, but do not have a 5 of 6 HLA-match sibling donor. Treatment may consist of:
  * Additional consolidation chemotherapy (3-4 cycles of cytarabine +/- an anthracycline agent, or other consolidation)
  * Autologous transplantation
  * Non-Myeloablative unrelated-donor transplant, +/- TLI and ATG conditioning
  * Umbilical cord blood transplantation
  * Haploidentical transplantation
  Best standard care: Intervention consist of:
  * Consolidation chemotherapy (3-4 cycles of cytarabine +/- an anthracycline agent, or other consolidation)
  * Autologous transplantation
  * Non-Myeloablative unrelated-donor transplant, +/- TLI and ATG conditioning
  * Umbilical cord blood transplantation
  * Haploidentical transplantation
Period: Overall Study
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Started | 25 | 33
Completed | 25 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care | Total
Number analyzed (Participants) | 25 | 33 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 26 | 46
  >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (5.1) | 60 (6) | 60 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 14 | 22 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 25 | 30 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 0 | 2 | 2
  White | 22 | 21 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 33 | 58

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time interval between the date of attaining a first complete remission (CR) and the date of death from any cause. The outcome is reported as the number of participants alive (without dispersion).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 33
Participants | 9 | 13

2. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival is defined as the time interval between the date of attaining a first complete remission (CR) and the date of relapse. Disease free survival (DFS) will compared to conventional therapy vs Non-myeloablative Host Conditioning (NMA HCT). The outcome is reported as the number of participants which never experienced disease relapse (without dispersion).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 33
Participants | 5 | 9

3. Secondary Outcome: Non-relapse Mortality
Description: Non-relapse mortality is defined as death that occurs after therapy, from any cause except a cause associated with relapse. This will be reported as the number of participants experiencing non-relapse mortality (a number without dispersion).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 33
Participants | 1 | 2

4. Secondary Outcome: Relapse Rate
Description: Relapse will be determined as ≥ 5% blast cells in the bone marrow, not secondary to regeneration after myelosuppressive therapy; OR emergence of extramedullary leukemia; OR the re-emergence of blasts in the peripheral blood. The outcome will be reported as the number and percentage of participants that meet these criteria (a number without dispersion).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 33
Participants | 20 | 24

5. Secondary Outcome: Transplant-related Mortality
Description: Transplant-related mortality will be assessed as any death occurring within 6 months post-transplant, from any cause except relapse. It will be measured at 100 day and 6 months after transplant. The outcome is expressed as at the number of participants experiencing transplant-related mortality (a number without dispersion).
Time Frame: 100 days and 6 months
Population: Participants in the Best Standard Care arm did not receive transplant, and are not evaluable for transplant outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 0
Participants
  At 100 days | 0 |
  At 6 months | 1 |

6. Secondary Outcome: Complete Donor Hematopoietic Cell Chimerism
Description: Complete donor hematopoietic cell chimerism was evaluated in transplant recipients. Complete donor chimerism will be assessed as the presence of > 95% donor T-cells (CD3+) in the blood. The outcome is reported as the percentage of participants that achieve complete donor chimerism, a number without dispersion.
Time Frame: 2 years
Population: Participants in the Best Standard Care arm did not receive transplant, and are not evaluable for transplant outcomes.
Measure: Number; unit: percentage of participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 0
percentage of participants | 56 |

7. Secondary Outcome: Early Graft Loss
Description: Early graft loss means a failure to achieve donor T-cell chimerism of > 5% at any time after transplant. The outcome is reported as the percentage of participants that experience early graft loss, a number without dispersion.
Time Frame: 2 years
Population: Participants in the Best Standard Care arm did not receive transplant, and are not evaluable for transplant outcomes.
Measure: Number; unit: percentage of participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 0
percentage of participants | 4 |

8. Secondary Outcome: Patients Completing the Intended Therapy in Both Arms
Description: The assessment for completion of the intended therapy (in both arms) will be reported as the percentage of participants, a number without dispersion
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
Number analyzed (Participants) | 25 | 33
percentage of participants | 100 | 81.8

ADVERSE EVENTS:
Time Frame: 2 years
Description: Non-serious adverse events were not collected in this study.
Arm/Group | Allo-HSCT + TLI + ATG | Best Standard Care
All-Cause Mortality (participants affected / at risk) | 16/25 | 20/33
Serious Adverse Events (participants affected / at risk) | 20/25 | 24/33
Other Adverse Events (participants affected / at risk) | 0/25 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allo-HSCT + TLI + ATG (N=25) | Best Standard Care (N=33)
Relapse, leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 (20) | 24 (24)
Death not otherwise specified (General disorders) | 1 (1) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No